CLINICAL TRIAL: NCT01863017
Title: Pilot Study of Startle-response Test to Assess Transcranial Direct Current Stimulation- Induced Modulation of Hyperphagia in Prader-Willi Syndrome
Brief Title: Pilot Study of Startle-response Test to Assess Transcranial Direct Current Stimulation-induced Modulation of Hyperphagia in Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Prader-Willi Syndrome Association USA (Other); Harvard Medical School (HMS and HSDM) (Other); Foundation for Prader-Willi Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13155
Record Dates: First submitted 2013-04-30; First posted 2013-05-27 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Hyperphagia; Prader-Willi Syndrome
Keywords: Obesity; Over weight
MeSH Terms: conditions — Hyperphagia; Prader-Willi Syndrome; Obesity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham tDCS (Sham Comparator): Five consecutive sessions of no tDCS. Each session will last approximately 30 minutes. Current will be applied for 20 minutes. Less than 3 minutes of tDCS has been shown to induce no lasting effects. Normal weight control participants will receive one sham session and one active session.
  Interventions: Device: tDCS
- Active tDCS (Experimental): Five consecutive sessions of tDCS administered. Each session will take about 30 minutes. Normal weight control participants will receive one sham session and one active session.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS
  Other Names: ActivaDoseII

SUMMARY:
The purpose of this study is to determine the effects of transcranial direct current stimulation (tDCS) as it modifies hyperphagia in obese subjects, non-obese subjects, and subjects with Prader-Willi syndrome (PWS).

DETAILED DESCRIPTION:
PWS is characterized by hypotonia, feeding difficulties, developmental delay and failure to thrive during infancy, and by an insatiable appetite (hyperphagia), rapid weight gain and obesity in early childhood.

Hyperphagia is one of the most prominent and debilitating features of PWS, and currently no pharmaceutical drug has been successful in decreasing appetite in such patients.

tDCS is a safe, noninvasive method whereby a weak electric current is directly transmitted into the brain via external electrodes connected to a 9-volt radio battery. It is based on decades-old observations that nerve cell firing can be altered by low amplitude direct current (DC). The researchers in this study believe that tDCS may have a positive impact on hyperphagia and weight.

In this study, the investigators intend to assess whether the effects tDCS differ between obese subjects, non-obese subjects, and subjects with Prader-Willi syndrome by measuring the amplitude and latency of eyeblink startle responses to a set of food- and non-food-related visual stimuli in all subjects, various hyperphagia questionnaires, and cognitive and behavioral assessments. It is hypothesized that as a group, subjects with Prader-Willi syndrome will demonstrate behavioral and psychometric evidence of abnormal food image processing, craving and associated behaviors relative to our control groups, and this group may receive potentially beneficial effects from tDCS sessions. Obese subjects are also predicted to have decreased hyperphagia and food cravings as a result of tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals and individuals diagnosed with Prader-Willi syndrome
* Provide informed consent to participate in the study
* Body Mass Index (BMI) <25kg/m2 (for non-obese subjects only)
* Body Mass Index (BMI) ≥30kg/m2 (for obese subjects only)

Exclusion Criteria:

* Subject is pregnant at time of enrollment in the study.
* Contraindications to tDCS:

  1. metal in the head
  2. implanted brain medical devices
* Clinically significant and unstable medical disorders (e.g., uncontrolled diabetes, uncompensated cardiac issues, heart failure, pulmonary issues, or chronic obstructive pulmonary disease) as self-reported.
* Clinically significant and unstable psychiatric disorders (e.g., schizophrenia, schizoaffective disorder, other psychosis, bipolar illness, severe depression) as self-reported.
* Significant visual impairment, as self-reported
* History of auditory deficiencies, as self-reported
* History of alcohol or substance abuse within the last 6 months as self-reported
* Use of carbamazepine within the past 6 months as self-reported.
* Current use of antidepressants
* History of neurological disorders as self-reported
* History of neurosurgery as self-reported

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10-06 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merlin G. Butler, MD, PhD, Principal Investigator — University of Kansas Medical Center; Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Prader-Willi Homes of Oconomowoc, Dousman, Wisconsin

REFERENCES:
- [Background] Bravo GL, Poje AB, Perissinotti I, Marcondes BF, Villamar MF, Manzardo AM, Luque L, LePage JF, Stafford D, Fregni F, Butler MG. Transcranial direct current stimulation reduces food-craving and measures of hyperphagia behavior in participants with Prader-Willi syndrome. Am J Med Genet B Neuropsychiatr Genet. 2016 Mar;171B(2):266-75. doi: 10.1002/ajmg.b.32401. Epub 2015 Nov 21. PMID 26590516

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tDCS: Five consecutive sessions of no transcranial direct current stimulation (tDCS). Each session will last approximately 30 minutes. Current will be applied for 20 minutes. Less than 3 minutes of tDCS has been shown to induce no lasting effects. Normal weight control participants will receive one sham session and one active session.
  tDCS
- Active tDCS: Five consecutive sessions of tDCS administered. Each session will take about 30 minutes. Normal weight control participants will receive one sham session and one active session.
  tDCS
Period: Overall Study
Arm/Group | Sham tDCS | Active tDCS
Started | 12 | 19
Normal Weight Participants | 5 | 5
Obese Participants | 4 | 7
Participants With PWS (Prader-Willi syndrome (PWS)) | 3 | 7
Completed | 12 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham tDCS: Five consecutive sessions of no tDCS. Each session will last approximately 30 minutes. Current will be applied for 20 minutes. Less than 3 minutes of tDCS has been shown to induce no lasting effects. Normal weight control participants will receive one sham session and one active session.
  tDCS
- Total: Total of all reporting groups
Arm/Group | Sham tDCS | Active tDCS | Total
Number analyzed (Participants) | 12 | 19 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 19 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at baseline was collected for all adult participants
  years
    all patients | 33.2 (13.7) | 39.3 (13.6) | 35.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 12 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Amplitude of Eyeblink Startle Responses
Description: Muscle contractions generated by the orbicularis oculi were recorded by a BIOPAC systems bioamplifier (model EMG 100c) passing 10-500 Hz signals, sampling at a rate of 2000/second and amplified by a factor of 5000. Eyeblink startle-responses were measured in response to food and non-food images at two lead-intervals (2500 ms and 6000 ms) to assess emotional responses (e.g., early and late, respectively) for each picture stimulus. Startle responses were assessed during (e.g., while viewing the food, puppy, etc.) and between (e.g., during washout periods; no-images) visual image-processing. Omnibus amplitudes are presented for sham vs active treatment groups for all participants, individuals with obesity and Prader Willi syndrome relative to lean controls.
Time Frame: Amplitude of Eyeblink Startle at Day 30 relative to normal weight controls
Population: All participants
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 12 | 19
microvolts
  All Participants | 0.006 (0.001) | 0.001 (0.001)
  Obese Participants: number analyzed (Participants) | 4 | 7
  Obese Participants | 0.008 (0.002) | 0.001 (0.001)
  Participants with PWS: number analyzed (Participants) | 3 | 7
  Participants with PWS | 0.004 (0.002) | 0.001 (0.001)

2. Primary Outcome: Dykens Hyperphagia Questionnaire
Description: The Dykens Hyperphagia Questionnaire is a 13-item instrument that was specifically designed to measure food-related preoccupations and problems, as well as the severity of these concerns. Items on the questionnaire are rated on a five-point scale (1: not a problem to 5: severe and/or frequent problem). Possible scores on the questionnaire range from a minimum score of 0 to a maximum score of 65. Higher scores indicate greater hyperphagia.
Time Frame: Total Score Day 30
Population: all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 12 | 19
score on a scale
  Normal Weight Participants: number analyzed (Participants) | 5 | 5
  Normal Weight Participants | 19.8 (4.0) | 22.1 (6.7)
  Obese Participants: number analyzed (Participants) | 4 | 7
  Obese Participants | 15.3 (5.1) | 24.8 (5.1)
  Participants with PWS: number analyzed (Participants) | 3 | 7
  Participants with PWS | 28.3 (6.1) | 25.3 (6.0)

3. Secondary Outcome: Three-Factor Eating Questionnaire
Description: The Three-Factor Eating Questionnaire is a self-completed, 51-item questionnaire that measures both cognitive and behavioral aspects of eating (dietary restraint, disinhibition, and hunger), and comprises two parts. Part 1 includes 36 true/false questions, and part 2 includes 14 questions on a four point Likert scale (1= rarely, 2 = sometimes, 3 = usually, 4 = always) and 1 question on a five point Likert scale (1 = eat whatever you want, whenever you want it to 5 = constantly limiting food intake, never 'giving in'; other questions). Higher scores indicate more severe pathology.
Time Frame: Total Scores at Day 30
Population: All participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 12 | 19
score on a scale
  Normal Weight Participants: number analyzed (Participants) | 5 | 5
  Normal Weight Participants | 19.82 (9.1) | 20.5 (10.3)
  Obese Participants: number analyzed (Participants) | 4 | 7
  Obese Participants | 16.3 (8.0) | 25.1 (10.7)
  Participants with PWS: number analyzed (Participants) | 3 | 7
  Participants with PWS | 32.7 (5.9) | 27.8 (5.0)

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Sham tDCS: Brief Stimulation
- Active tDCS: Transcranial Direct Current Stimulation for 30 minutes
Arm/Group | Sham tDCS | Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/19
Other Adverse Events (participants affected / at risk) | 0/12 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No